CLINICAL TRIAL: NCT01360112
Title: Malaria Transmission Blocking Assay Development and Gametocyte Carriage in a Vaccine Testing Site in Mali
Brief Title: Preventing the Spread of Malaria in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911143; 11-I-N143
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2017-11-16

CONDITIONS: Malaria
Keywords: Mosquito; Membrane; Feeding; Parasites; Infection; Malaria
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A vaccine which interrupts malaria transmission is a critical tool to achieve the ultimate goal of eradication of this disease. Transmission blocking vaccines work by inducing antibody in vaccinated individuals that inhibits the development of malaria parasites in the mosquito, thus interrupting the cycle of transmission to the next human host. Efficacy of these vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory strain mosquitoes, but these assays need to be qualified to determine to what extent they are predictive of transmission blocking in the field. Clinical trials of transmission blocking vaccines are also anticipated and have started in this community. This protocol will use a nested casecontrol cohort design to compare results of mosquito feeding assays in a malaria exposed population in Bancoumana and surrounding villages in Mali. Households will be identified using census data and individuals will be consented for participation. Malaria smears will be obtained at monthly visits, and gametocytemic individuals will be asked to participate in direct feed experiments using insectary-raised mosquitoes. Infectivity in these mosquitoes will be compared against those of mosquitoes fed in membrane feeding assays in Mali and the USA. Data will also be obtained on gametocyte and parasite carriage rates through the year. A total of 250 volunteers from Bancoumana, ages 3 months to 50 years, were initially enrolled in 2011. In 2012, an additional 250 adults from Bancoumana were enrolled and participants older than 5 years of age who were enrolled in 2011 and wanted to continue participation were re-enrolled into the study. A transmission blocking vaccine trial started in May 2013, and has enrolled participants from this adult cohort in that study. Up to 50 new adults from Bancoumana and surrounding villages will be enrolled in 2014 and those volunteers previously enrolled into the study over theage of 5 years old will be offered re-enrollment into the study.

DETAILED DESCRIPTION:
A vaccine which interrupts malaria transmission is a critical tool to achieve the ultimate goal of eradication of this disease. Transmission blocking vaccines work by inducing antibody in vaccinated individuals that inhibits the development of malaria parasites in the mosquito, thus interrupting the cycle of transmission to the next human host. Efficacy of these vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory strain mosquitoes, but these assays need to be qualified to determine to what extent they are predictive of transmission blocking in the field. Clinical trials of transmission blocking vaccines are also anticipated and have started in this community. This protocol will use a nested casecontrol cohort design to compare results of mosquito feeding assays in a malaria exposed population in Bancoumana and surrounding villages in Mali. Households will be identified using census data and individuals will be consented for participation. Malaria smears will be obtained at monthly visits, and gametocytemic individuals will be asked to participate in direct feed experiments using insectary-raised mosquitoes. Infectivity in these mosquitoes will be compared against those of mosquitoes fed in membrane feeding assays in Mali and the USA. Data will also be obtained on gametocyte and parasite carriage rates through the year. A total of 250 volunteers from Bancoumana, ages 3 months to 50 years, were initially enrolled in 2011. In 2012, an additional 250 adults from Bancoumana were enrolled and participants older than 5 years of age who were enrolled in 2011 and wanted to continue participation were re-enrolled into the study. A transmission blocking vaccine trial started in May 2013, and has enrolled participants from this adult cohort in that study. Up to 50 new adults from Bancoumana and surrounding villages will be enrolled in 2014 and those volunteers previously enrolled into the study over theage of 5 years old will be offered re-enrollment into the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a volunteer to participate in the study:

1. Age between 3 months and 50 years, inclusive
2. Good general health as a result of review of medical history and/or clinical testing at the time of screening
3. Available for the duration of the study (1 year)
4. Willingness to participate in the study as evidenced by signing the informed consent document, or by fingerprinting the consent document with the signature of a witness
5. Known resident of the village of the study
6. Willingness to allow stored laboratory specimens to be used for future research.
7. In addition to the above criteria, the expanded adult cohort must be willing to consider participation in a future malaria vaccine trial.

EXCLUSION CRITERIA:

A volunteer will be excluded from participating in this study if any one of the following criteria is fulfilled:

1. Pregnancy as determined by history or a positive urine Beta-hCG test at any point during the study.
2. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
3. Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
4. Participation in another investigational vaccine or drug trial while this study is ongoing.
5. Previous receipt of experimental malaria vaccine.
6. Baseline hemoglobin < 8.5 g/dL

   In addition to above criteria, a volunteer will be excluded from participating in the transmission blocking assay part of the study if the following criteria is fulfilled:
7. History of reactions to mosquito bites with severe itching or swelling, or lasting longer than 3 days

Ages: 3 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 816 (Actual)
Dates: Start 2011-05-20; Study Completion 2017-11-16

PRIMARY OUTCOMES:
a) Mosquito infectivity by DF, DMFA (a, b, and c), and SMFA (d and e), as measured by infection rate (number of infected vs. un- nfected mosquitoes), and oocyst counts in infected mosquitoes, both determined using microscopy. | 24 months
b) The period prevalence and density of gametocytes throughout the study period, as detected by thick smear and nucleic acid based techniques | 24 months

SECONDARY OUTCOMES:
a)Antibody levels to sexual P. falciparum antigens, and other antigens of interest. | 24 months
b)Mosquito infectivity as measured by circumsporozoite protein (CSP) ELISA. | 24 months
c)Hemoglobin level as measured by HemoCue. | 24 months
d)Hemoglobin variants (hemoglobin S, C, alpha thalassemia), G6PD status, blood group/Rh. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Cheru L, Wu Y, Diouf A, Moretz SE, Muratova OV, Song G, Fay MP, Miller LH, Long CA, Miura K. The IC(50) of anti-Pfs25 antibody in membrane-feeding assay varies among species. Vaccine. 2010 Jun 17;28(27):4423-9. doi: 10.1016/j.vaccine.2010.04.036. Epub 2010 Apr 29. PMID 20434549
- [Background] Birkett AJ. PATH Malaria Vaccine Initiative (MVI): perspectives on the status of malaria vaccine development. Hum Vaccin. 2010 Jan;6(1):139-45. doi: 10.4161/hv.6.1.10462. Epub 2010 Jan 29. No abstract available. PMID 20009524
- [Background] Diallo M, Toure AM, Traore SF, Niare O, Kassambara L, Konare A, Coulibaly M, Bagayogo M, Beier JC, Sakai RK, Toure YT, Doumbo OK. Evaluation and optimization of membrane feeding compared to direct feeding as an assay for infectivity. Malar J. 2008 Dec 2;7:248. doi: 10.1186/1475-2875-7-248. PMID 19055715